CLINICAL TRIAL: NCT05382702
Title: Fear, Gastrointestinal Distress, and Interoception: Physiological and Psychological Mechanisms in Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio University (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 21-F-14; R15MH128703 (NIH)
Record Dates: First submitted 2022-05-11; First posted 2022-05-19 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Feeding and Eating Disorders
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Fat Yogurt - Low Fat Yogurt (Other): Participants will eat yogurt described as 'high fat' at Study Visit 2 and yogurt described as 'low fat' at Study Visit 3.
  Interventions: Other: Test meal description changed
- Low Fat Yogurt - High Fat Yogurt (Other): Participants will eat yogurt described as 'low fat' at Study Visit 2 and yogurt described as 'high fat' at Study Visit 3.
  Interventions: Other: Test meal description changed

INTERVENTIONS:
Other: Test meal description changed — Using a within-subjects crossover design, on two separate mornings participants will eat yogurt described as 'high fat' and 'low fat.' In actuality, the meals will not differ.

SUMMARY:
The proposed study tests fear, gut peptide response, and perceptions of fullness as causes of gastrointestinal distress and eating disorder maintenance.

ELIGIBILITY:
Inclusion Criteria:

* female
* DSM-5 eating disorder
* score 16 or higher on the Clinical Impairment Assessment
* experience nausea or stomachache after eating at least "sometimes"
* 18 to 40 years old
* body mass index between 18.5 and 26.5 kg/m2

Exclusion Criteria:

* medical conditions affect appetite or weight
* Recent pregnancy or current breastfeeding
* Dairy, strawberry or honey food allergy
* Specific phobia, blood-injection-injury type

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 152 (Estimated)
Dates: Start 2022-04-22 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Subjective rating of fear | -10 minutes, 0 minutes (immediately after the intervention), and 10 minutes post-intervention
  Area under the curve with respect to increase (AUCi) from the 10 minutes period prior to the meal until immediately after the meal will be used to characterize changes in Visual Analogue Scale ratings of momentary fear ranging from "Not at All" to "Extreme." Subjective fear immediately before the meal will be used in mediation models.
Skin conductance | -10 minutes, 0 minutes (immediately after the intervention), and 10 minutes post-intervention
  Skin conductance data will be collected using a Biopac Bionomadix EDA System. Difference scores will be computed for both test meals by comparing mean skin conductance level (expressed in log units) over the 10 minute meal period to the 10 minute period before the meal.
Gastrointestinal distress | -10 minutes, 0 minutes (immediately after the intervention), 10 minutes, 20 minutes, 30 minutes, 60 minutes and 90 minutes post-intervention
  Gastrointestinal distress will be the averaged visual analogue scale ratings of "Nausea" and "Stomach Ache" ranging from "Not At All" to "Extreme." Area under the curve with respect to increase (AUCi) from the 10 minutes period prior to the meal until immediately after the meal will be used to characterize changes gastrointestinal distress. The 20-minute assessment of gastrointestinal distress will be used for the hypothesis testing mediators of the relationship between fear and gastrointestinal distress and the 30 minute assessment will be used for the exploratory serial multiple mediation model.
Cholecystokinin response | 0 minutes (immediately after the intervention), 10 minutes, 20 minutes, 30 minutes, 60 minutes and 90 minutes post-intervention
  Blood will be drawn repeatedly. Cholecystokinin (CCK) values in plasma will be quantified using a commercially available enzyme immunoassay. Area under the curve with respect to increase (AUCi) will be calculated for all time periods to compare between test meal instructions. CCK values 10 minutes after the intervention will be used in mediation models.
Peptide YY response | 0 minutes (immediately after the intervention), 10 minutes, 20 minutes, 30 minutes, 60 minutes and 90 minutes post-intervention
  Blood will be drawn repeatedly. PYY3-36 values in plasma will be quantified using a commercially available enzyme immunoassay. Area under the curve with respect to increase (AUCi) will be calculated for all time periods to compare between test meal instructions. PYY values 10 minutes after the intervention will be used in mediation models.
Subjective rating of fullness | 0 minutes (immediately after the intervention), 10 minutes, 20 minutes, 30 minutes, 60 minutes and 90 minutes post-intervention
  Fullness will be the averaged visual analogue scale ratings of "full" and "satiated(satisfied)" ranging from "Not At All" to "Extreme." Area under the curve with respect to increase (AUCi) will be used to characterize changes in fullness from immediately before the test meal to 90 minutes after. The 10-minute assessment of fullness will be used in testing fullness as a mediator of the relationship between fear and gastrointestinal distress and the 20 minute assessment will be used for the exploratory serial mediation model.
Urges to restrict food intake | 60 minutes post-intervention
  Visual analogue scales will assess momentary "urge to restrict" from "Not At All" (0) to "Extreme" (100). The 60 minute assessment will be used for the exploratory serial mediation model.

CONTACTS AND LOCATIONS:
Overall Officials: Katherine J Forney, PhD, Principal Investigator — Ohio University
Locations (1):
- Ohio University, Athens, Ohio, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared according to the NIMH Data Sharing Policy (NOT-MH-19-033), including being shared with the NIMH Data Archive.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2022-04-27): https://cdn.clinicaltrials.gov/large-docs/02/NCT05382702/Prot_SAP_000.pdf
  • Informed Consent Form: Online Screen (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT05382702/ICF_007.pdf
  • Informed Consent Form: In Person Consent (2024-12-02): https://cdn.clinicaltrials.gov/large-docs/02/NCT05382702/ICF_008.pdf